CLINICAL TRIAL: NCT06433245
Title: Outcome Following Use of Different Concentrations of Sodium Hypochlorite as Wound Lavage and Hemostatic Agent in Partial Pulpotomy: A Randomised Control Trial
Brief Title: Outcome Following Use of Different Concentrations of NaOCl as Wound Lavage and Hemostatic Agent in Partial Pulpotomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Ridhi Karwal
Record Dates: First submitted 2024-05-22; First posted 2024-05-29 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Irreversible Pulpitis; Extremely Deep Caries; Partial Pulpotomy
Keywords: partial pulpotomy; sodium hypochlorite; mature permanent mandibular molars; hemostatic agent

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The operator, patient and the outcome assessor will be masked to the group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control: 3% sodium hypochlorite (Active Comparator): After partial pulpotomy procedure, pulp wound will be irrigated with 3% sodium hypochlorite and haemostasis will be achieved by placing the cotton pellet soaked with 3% sodium hypochlorite on the amputated pulp.
  Interventions: Procedure: effect of 3% and 5% sodium hypochlorite on outcome of partial pulpotomy in teeth with clinical signs indicative of irreversible pulpitis.
- Test: 5% sodium hypochlorite (Experimental): After partial pulpotomy procedure, pulp wound will be irrigated with 5% sodium hypochlorite and haemostasis will be achieved by placing the cotton pellet soaked with 5% sodium hypochlorite on the amputated pulp.
  Interventions: Procedure: effect of 3% and 5% sodium hypochlorite on outcome of partial pulpotomy in teeth with clinical signs indicative of irreversible pulpitis.

INTERVENTIONS:
Procedure: effect of 3% and 5% sodium hypochlorite on outcome of partial pulpotomy in teeth with clinical signs indicative of irreversible pulpitis. — After caries removal and pulp exposure pulp tissue is amputated and hemostasis is achieved with 3% sodium hypochlorite in control group and 5% sodium hypochlorite in experimental group followed by capping with 2-3mm layer of MTA. A layer of RMGIC will be placed over the MTA. Then the tooth will be permanently restored with composite resin.

SUMMARY:
The aim of this randomised control trial is to compare the effect of different concentrations of NaOCl on outcome of partial pulpotomy in teeth with clinical signs indicative of irreversible pulpitis.

The main question it aims to answer are:

1. clinical and radiographic outcome of partial pulpotomy following use of 5% and 3% NaOCl in mature permanent teeth with clinical signs indicative of irreversible pulpitis.
2. OHRQoL and pain experience after use of 5% and 3% NaOCl during partial pulpotomy in teeth with clinical signs indicative of irreversible pulpitis.

DETAILED DESCRIPTION:
TITLE :- Outcome following use of different concentrations of NaOCl as wound lavage and hemostatic agent in partial pulpotomy: A Randomised control trial.

Question it aims to answer:

Does pulpal lavage using 3% and 5% sodium hypochlorite have comparable effect on outcome of partial pulpotomy in mature permanent teeth with clinical signs of irreversible pulpitis? P (Population) -Mature permanent mandibular molars with signs of irreversible pulpitis.

I (Intervention) - 5% NaOCl C (Comparison) - 3% NaOCl O (Outcome) - 1. Assessment of clinical and radiographic success at 12 months of follow up.

2. Assessment of OHRQoL and pain experience at baseline, post-operatively every 24 hours for 1 week and OHRQoL at 6 and 12 months.

In literature pertaining to vital pulp therapy procedures, there is often a focus on comparing various materials or treatment methodologies. However, the use of sodium hypochlorite, holds significant importance in ensuring the successful outcome of the procedure. The previous studies indicate that the use of NaOCl presents as a confounding factor, compounded by variations among operators in their choice of high and low concentrations of NaOCl.So, there is a pressing need for a direct comparative analysis to assess the influence of varying sodium hypochlorite concentrations on the overall efficacy and success rates of vital pulp therapy procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Mature permanent mandibular molars.
2. Teeth with clinical diagnosis of symptomatic irreversible pulpitis
3. Patients having normal periapical status with periapical index (PAI) score ≤ 2
4. Periodontally healthy teeth
5. Patients having physical status of class 1 or 2 according to ASA classification
6. Pulpal bleeding can be controlled within 6 minutes.
7. Presence of extremely deep carious lesion on radiograph -

Exclusion Criteria:

1) Non restorable teeth 2) Necrotic pulp evident upon exposure 3) Negative response to vitality test 4) Presence of sinus tract 5) Presence of soft tissue swelling 6) Radiographic signs of internal or external root resorption 7) Pregnant women

-

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 116 (Estimated)
Dates: Start 2024-05-23 (Actual); Primary Completion 2025-12-23 (Estimated); Study Completion 2025-12-23 (Estimated)

PRIMARY OUTCOMES:
Clinical success rate | baseline to 12 months
  Clinical criteria of success:-
  1. No pain or discomfort except for the first few days after treatment.
  2. No tenderness to palpation or percussion and the tooth is functional.
  3. Normal mobility and probing pocket depth.
  4. Healthy soft tissues around teeth with no swelling, sinus tract.
Radiographic success rate | Baseline to 12 months
  Radiographic success criteria:-
  1. No pathosis such as root resorption, furcal pathosis or new periapical pathosis evident on the radiograph.
  2. Complete radiographic healing

SECONDARY OUTCOMES:
Post Operative Pain | Baseline to 7 days
  To assess incidence and intensity of pain postoperatively at every 24 hours till 7 days using Visual analogue Scale of 0 to 100 millimeter line. Score 0 means no pain and Score100 means maximum pain. To assess incidence and intensity of pain postoperatively at every 24 hours till 7 days using Visual analogue Scale of 0 to 100 millimeter line. Score 0 means no pain and Score 100 means maximum pain
OHRQoL assessment | baseline and at 24 h, 2, 3, 4, 5, 6 and 7 days after the treatment, and then at 6 and 12 months.
  OHIP-14 questionnare will be used to assess the quality of life.It consists of questionnaire in seven dimensions: functional limitation, physical pain, psychological discomfort, physical disability, psychological disability, social disability, and handicap. It will be scored using a Lickert scale:
  never=0; hardly ever=1; occasionally=2; fairly often=3; very often=4. Total score will be calculated ranging from 0-56, with higher score denoting the worst OHRQoL

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Sanjay Tewari, MDS, Study Director — PGIDS, Rohtak, Haryana 124001
Locations (1):
- PIGDS, Rohtak, Haryana, India